CLINICAL TRIAL: NCT00506376
Title: Simple Versus Radical Hysterectomy for Stage I Cervical Cancer: Preferences of Women at High-Risk for Developing Cervix Cancer vs. Women Diagnosed With Cervix Cancer
Brief Title: Simple Versus Radical Hysterectomy for Stage I Cervical Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID02-741
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Hysterectomy; Interview
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical Treatment Preferences: Assessment of patient's feelings toward risks associated with surgical treatment of cervical cancer.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview that will take about 20 minutes to complete.

SUMMARY:
The primary objective of this study is to assess the preferences (values and utilities) of women for complications and recurrences associated with the surgical treatment of cervical cancer. A secondary objective of this study is to compare the preferences of women at high-risk for developing cervix cancer with the preferences of women who have already been diagnosed with cervix cancer.

DETAILED DESCRIPTION:
You will be asked to undergo a face to face interview. During the interview, you will be asked questions about your values and feelings about your health status. You will be shown a "feeling thermometer" and asked to rate how your health condition makes you feel. You will also be asked to rate how some of the risks of treatment of cervix cancer make you feel. You will be shown a "chance board" and asked to consider some of the possible outcomes of the disease and possible risks associated with the treatment of cervix cancer. You will be asked to consider the likelihood of achieving certain outcomes and of developing certain side effects due to the disease and/or treatment. The interview will take place in a private room in the clinic and should take around 20 minutes to complete.

This is an investigational study. As many as 96 women will participate in this study. Up to 48 women who are at high risk of developing cervix cancer and up to 48 women who have been diagnosed with cervix cancer will participate. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are at least 18 years of age.
2. Women who speak English
3. Women presenting to the Colposcopy Clinic in the Gynecologic Oncology Clinic at M.D. Anderson Cancer Center OR women with an established diagnosis of either Stage IA2 or IB1 cervix cancer treated with radical hysterectomy 3-24 months prior to presenting to the Gynecologic Oncology

Exclusion Criteria:

1. Women who are not 18 years of age.
2. Women who are non-English speakers.
3. Women with a diagnosis of any type of cancer other than cervical cancer.
4. Women who are currently pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants at high-risk for cervical cancer and those already diagnosed with cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2003-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Preference Assessment | Baseline + Interview

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte C. Sun, DrPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org